CLINICAL TRIAL: NCT01148641
Title: Acceptability of Lipid-based Nutrient Supplements (LNS) for Infants and Young Children in Guatemala
Brief Title: Acceptability of LNS for Infants and Young Children in Guatemala
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Other Study IDs: 201017829
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Malnutrition
Keywords: Lipid-based supplements; LNS; Acceptability; Infant nutrition; Guatemala; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LNS-regular: Lipid-based nutrient supplement, regular (peanut) flavor
  Interventions: Dietary Supplement: LNS
- LNS-cinnamon: Lipid-based nutrient supplement, cinnamon flavor
  Interventions: Dietary Supplement: LNS

INTERVENTIONS:
Dietary Supplement: LNS — Infants and young children will receive 10 g of LNS for test trial during 3 consecutive days (crossover design) and thereafter, 20 g per day for 14 days.
  Other Names: Lipid-based nutrient supplement

SUMMARY:
This study aims to assess the acceptability of lipid-based nutrient supplements (LNS) for use as nutritional supplements for infants and young children in Guatemala.

The study was conducted in three phases. Phase 1 was a test-feeding to compare the acceptability of two different flavors of LNS (peanut and cinnamon) in infants and young children and their mothers or caregivers in terms of taste, smell and texture, as well as amount of the test-dose consumed. In Phase 2, children in the Phase 1 trial received a 2-week supply of one of the LNS products, which they consumed daily in their homes for 14 days under real-life conditions. Direct observation of supplement use and in-depth interviews with mothers, caregivers and health staff providing services in communities will be part of this phase too. In Phase 3, focus group discussions (FGD) were held with participants (mothers and caregivers) as well as with health staff providing services in communities to discuss different aspects of infant and child feeding and best ways for the LNS product to be used in the context of Guatemala.

We hypothesized that both flavors of LNS would be accepted by Guatemalan infants and young children children and their mothers or caregivers.

DETAILED DESCRIPTION:
The study was carried out in two communities in the Suchitepéquez Department in partnership with Funcafé, a NGO subcontracted by the Ministry of Health (MOH) to implement the Programa de Extension de Cobertura (PEC) in Suchitepéquez. PEC provides basic medical care in remote communities that have limited access to MOH's health centers. This acceptability study was conducted in communities where PEC was implemented by Funcafé.

The children were randomly selected from a list of beneficiaries of PEC served by Funcafé and invited to participate. Eligibility for participation in the study was determined at the time of recruitment in the homes of potential participants, by administration of a screening questionnaire by study staff.

All caregivers who completed the home use trial were invited to participate in the FGD. Funcafé staff members (i.e. Institutional facilitators, Community facilitators and Community monitors) were randomly selected from the employee roster and potential participants were invited to participate in FGD using a standard recruitment script.

The study was approved by the IRB of the University of California, Davis. Unawareness of whether a child was intolerant of peanut or milk products did not prevent participation, but the child was provided with a small dose of LNS (~5 g) and asked to remain under observation by study staff for at least one hour. After this initial test, caregivers were also given the project's mobile phone number to call in case there were any symptoms during the next few hours. No allergic reactions or other adverse effects were observed or reported in any subject.

During the Test-feeding trial, the order of the versions of LNS tested was randomly determined for each subject. At the first home visit after recruitment (Day 0), the primary caregivers of the children were given an orientation about LNS. During the orientation, background data (e.g., socioeconomic and demographic information) were collected using a structured questionnaire and the experimental procedures were practiced, including initial tasting of the LNS mixed with food and completion of the tasting questionnaire, but no data on amount consumed or organoleptic preferences were recorded. The second home visit was Test Day 1, during which the actual tasting was recorded. All children were apparently healthy and had not eaten any food (including breast milk) during the previous hour, but during that time water was allowed. Caregivers were asked to provide 40 g (~3 tablespoons) of the complementary food they usually give to their children that was available at home, to which 10 g (~2 teaspoons) of LNS were mixed. The mother/caregiver of the child was asked to consume one teaspoon of the LNS + food mixture (~ 5 g), and then to feed the rest (~ 45 g) to the child after the mixture was re-weighed. The mother or caretaker rated the mixture's color, aroma, flavor and consistency based on her own opinion, and her perception of the infant's degree of liking using a 5-point pictorial hedonic scale (i.e., dislike very much, dislike, neutral, like, like very much). In order to test the different flavored LNS a third home visit was conducted (Test Day 2). The same procedures described above for Test Day 1 were followed on Day 2, but each child tasted the other LNS flavor. No overall or organoleptic (i.e., color, odor, taste and consistency) preferences were assessed on Day 2. Thus, total participation in this phase lasted 3 days, including the initial orientation day. At each test-feeding day, we collected data on infant's health (i.e., nasal discharge, cough, difficulty breathing, fever, diarrhea, vomit/nausea, ear infection, and any other symptom) and any possible reaction to the test meal.

For the Home use trial, primary caregivers of children who participated in the test-feeding trial received a two-week supply of LNS, which they were asked to add to their infants' prepared food each day. The daily ration of LNS was 20 g/day, provided in two 10-g sachets. In order to avoid bias, the LNS flavor to be distributed during the home-use trial was randomly assigned without taking into account the child's preference (if any) as explained above. To ensure that subjects consumed the entire daily ration, caregivers were instructed, to mix each sachet with 2-3 tablespoons of the home-prepared food, to be fed to the child before the rest of the food was offered.

After the end of the first week of supplementation, a field worker visited the household of each participant to count the empty (used) sachets and ask questions about any child illness. At the end of two weeks, a field worker visited each participant in his/her home to repeat the morbidity questionnaire and conduct an exit interview with the mother/caregiver to assess their perceptions, use and possible intra-household distribution of the product, ease/difficulty of providing the supplement 2 times/day, and foods used to mix with the supplement.

In addition, open ended questions were asked at the exit interview to explore the caregivers' views about important characteristics of foods appropriate for infants and young children, opportunities and barriers to using a nutrient supplement "just for children of a certain age" in the family, perceptions of the use of LNS for children, and recognition of the problem of malnutrition in their communities.

The FGD were led by an experienced focus group facilitator, assisted by a note-taker who audio-recorded the discussions and took notes on group dynamics and non-verbal interactions between participants. Each focus group included 8-10 participants, and lasted for approximately 60-90 minutes.

Four FGD (two per community) were conducted with primary caregivers of the children who had consumed LNS during the test-feeding and the home-use trial. The main purpose of the FGD was to get input on appropriate supplement names and packaging designs for the LNS product in Guatemala, flavors appropriate for infants and young children, and appropriate messages for promotion of LNS for children. A brainstorming approach was used to explore possible names for the supplement, followed by secret vote to short list the names based on participants' preferences. Exploration of ideas about packaging designs started with drawings which were then organized by theme. A discussion to generate consensus on the key elements that the label should include was facilitated. A group design for the packaging was the final product of FGD.

The main objective of the FGD with Funcafé personnel was to elicit their opinion on how the LNS could be incorporated into Funcafé's program operation.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-18 months of age.
* Consuming solid foods for at least the past 30 days.
* Apparently healthy and not presently suffering from an acute illness (e.g., fever, diarrhea, acute respiratory tract infection).
* No known allergy to peanuts or other food products (as reported on the screening questionnaire by the mother/primary caregiver).
* Not severely malnourished [mid-upper arm circumference (MUAC) > 115 mm].
* Maternal/caregiver willingness to feed the infant with LNS over a maximum 3 test days, and over the 2 week home-use period, and report on his/her consumption and reactions and practices for daily use. Willingness to participate in discussion groups.
* Planning to remain in study area for at least the following three weeks.

Exclusion Criteria:

* Children under 6 months of age.
* All subjects with known peanut, soy or milk allergies.
* In poor health or ill at the time of recruitment.
* Severely malnourished children [mid-upper arm circumference (MUAC) < 115 mm].
* Not willing to participate in study procedures.
* Leaving the study area in the following three weeks.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: - Children 6-18 months of age.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
amount of LNS consumed | 2 weeks
  Amount of LNS consumed in the test trial in grams
time of consumption | 2 weeks
  Avg how long it takes to eat the LNS mins
amount of LNS sachets consumed in the home-use trial | 2 weeks
  # of sachets consumed

SECONDARY OUTCOMES:
qualitative assessment of mothers and caregivers opinions | 2 weeks
  Focus group discussion (qualitative results) discuss different aspects of infant and child feeding and best ways for the LNS product to be used in the context of Guatemala.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G Dewey, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Fundacion de la Caficultura para el Dessarrollo Rural (FUNCAFE), Mazatenango, Departamento de Suchitepéquez, Guatemala